CLINICAL TRIAL: NCT02422927
Title: Effect of a Nutraceutical Combination on Endothelial Injury and C-reactive Protein in Patients With Low-grade Systemic Inflammation
Brief Title: Nutraceutical Combination in Patients With Low-grade Systemic Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Matteo Pirro, M.D., PhD, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPerugia01
Record Dates: First submitted 2015-04-13; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Atherosclerosis; Inflammation; Hypercholesterolemia
Keywords: C-Reactive Protein; Endothelial Microparticles; Endothelium; Nutraceutical; Cholesterol
MeSH Terms: conditions — Atherosclerosis; Inflammation; Hypercholesterolemia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care + Placebo (Placebo Comparator): low-cholesterol/low-saturated fat diet and a regular aerobic physical activity schedule + once daily placebo
  Interventions: Other: Standard of Care; Other: Placebo
- Nutraceutical combination (Active Comparator): low-cholesterol/low-saturated fat diet and a regular aerobic physical activity schedule + Nutraceutical combination
  Interventions: Dietary Supplement: Nutraceutical Combination; Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Nutraceutical Combination — red yeast rice extract 200 mg (equivalent to 3 mg monacolins), policosanol 10 mg, berberine 500 mg, 0.2 mg folic acid, coenzyme Q10 2 mg, and astaxanthin 0.5 mg once daily
  Other Names: Armolipid Plus, Rottapharm-Madaus
  Arms: Nutraceutical combination
Other: Standard of Care — low-cholesterol/low-saturated fat diet and regular aerobic physical activity schedule
Other: Placebo — placebo
  Arms: Standard of Care + Placebo

SUMMARY:
The investigators tested if a nutraceutical combination with red yeast rice, berberine and policosanol (NC) can significantly modify inflammation, lipid profile and markers of endothelial injury (endothelial microparticles) in subjects with elevated levels of high-sensitivity C-reactive protein (hsCRP).

DETAILED DESCRIPTION:
Will be included in the study 100 subjects with suboptimal LDL cholesterol levels (LDL 100-160 mg / dL) and hsCRP levels> 2 mg / L, divided into two groups of equal numbers, matched by by sex and age, randomized to receive a nutraceutical combination containing red yeast 200 mg, berberine 500 mg and policosanol 10 mg (NC) in combination with a low-cholesterol diet (<200 mg / day) or a low-cholesterol diet only (Standard of Care - SOC).

All subjects at the time of inclusion in the study protocol will be prescribed the SOC for a period of 30 days (Lipid Stabilization Period: LSP); After 30 days LSP it will be performed randomization in the two intervention arms: NC + SOC or SOC.

ELIGIBILITY:
Inclusion Criteria:

* LDL cholesterol <160 mg/dl (4,14 mmol/l);
* hsCRP >2 mg/L;

Exclusion Criteria:

* triglycerides >500 mg/dL (5.6 mmol/L);
* current or previous treatment with lipid-lowering drugs or with other drugs supposed to modify vascular damage and/or repair (antiplatelet, anti-hypertensive and antioxidant drugs);
* current or previous treatment with hormone replacement therapy for menopause vasomotor symptoms;
* evidence of liver dysfunction or alanine-aminotransferase (ALT) levels twice above the upper normal limit;
* creatin-kinase (CK) levels thrice above the upper normal limit
* history or clinical evidence of previous or current cardiovascular disease;
* presence of strong cardiovascular risk factors such as: serum creatinine levels >2 mg/dL, diabetes mellitus, uncontrolled systemic arterial hypertension (systolic blood pressure >190 mg/dL or diastolic blood pressure >100 mg/dL); history of cancer in the former 5 years before recruitment; not adequately treated hypothyroidism (TSH levels >1,5 times the upper normal limit);
* history of malignancy in the previous 5 years before screening;
* not adequately treated hypothyroidism (TSH levels >1,5 times the upper normal limit);
* previous or current alcohol or drugs abuse;
* history or clinical evidence of chronic inflammatory disease such as severe arthritis, systemic lupus erythematosus or chronic inflammatory bowel disease;
* current or previous use of immunosuppressant agents or long term glucocorticoids
* history or clinical evidence of any severe concomitant disease which may compromise subject's safety or its possibility to carry out the study.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in LDL cholesterol at 3 months | 3 months after treatment randomization

SECONDARY OUTCOMES:
Change from Baseline in Circulating endothelial microparticles at 3 months | 3 months after treatment randomization
Change from Baseline in C-reactive protein at 3 months | 3 months after treatment randomization

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Pirro, MD, PhD, Principal Investigator — University Of Perugia

REFERENCES:
- [Background] McGorrian C, Yusuf S, Islam S, Jung H, Rangarajan S, Avezum A, Prabhakaran D, Almahmeed W, Rumboldt Z, Budaj A, Dans AL, Gerstein HC, Teo K, Anand SS; INTERHEART Investigators. Estimating modifiable coronary heart disease risk in multiple regions of the world: the INTERHEART Modifiable Risk Score. Eur Heart J. 2011 Mar;32(5):581-9. doi: 10.1093/eurheartj/ehq448. Epub 2010 Dec 22. PMID 21177699
- [Background] Pirro M, Bergeron J, Dagenais GR, Bernard PM, Cantin B, Despres JP, Lamarche B. Age and duration of follow-up as modulators of the risk for ischemic heart disease associated with high plasma C-reactive protein levels in men. Arch Intern Med. 2001 Nov 12;161(20):2474-80. doi: 10.1001/archinte.161.20.2474. PMID 11700160
- [Background] Gerli R, Sherer Y, Vaudo G, Schillaci G, Gilburd B, Giordano A, Bocci EB, Allegrucci R, Marchesi S, Mannarino E, Shoenfeld Y. Early atherosclerosis in rheumatoid arthritis: effects of smoking on thickness of the carotid artery intima media. Ann N Y Acad Sci. 2005 Jun;1051:281-90. doi: 10.1196/annals.1361.069. PMID 16126969
- [Background] Gerli R, Vaudo G, Bocci EB, Schillaci G, Alunno A, Luccioli F, Hijazi R, Mannarino E, Shoenfeld Y. Functional impairment of the arterial wall in primary Sjogren's syndrome: combined action of immunologic and inflammatory factors. Arthritis Care Res (Hoboken). 2010 May;62(5):712-8. doi: 10.1002/acr.20117. PMID 20191479
- [Background] St-Pierre AC, Cantin B, Bergeron J, Pirro M, Dagenais GR, Despres JP, Lamarche B. Inflammatory markers and long-term risk of ischemic heart disease in men A 13-year follow-up of the Quebec Cardiovascular Study. Atherosclerosis. 2005 Oct;182(2):315-21. doi: 10.1016/j.atherosclerosis.2005.02.009. PMID 16159604
- [Background] Ridker PM, Rifai N, Clearfield M, Downs JR, Weis SE, Miles JS, Gotto AM Jr; Air Force/Texas Coronary Atherosclerosis Prevention Study Investigators. Measurement of C-reactive protein for the targeting of statin therapy in the primary prevention of acute coronary events. N Engl J Med. 2001 Jun 28;344(26):1959-65. doi: 10.1056/NEJM200106283442601. PMID 11430324
- [Background] Pirro M, Schillaci G, Paltriccia R, Bagaglia F, Menecali C, Mannarino MR, Capanni M, Velardi A, Mannarino E. Increased ratio of CD31+/CD42- microparticles to endothelial progenitors as a novel marker of atherosclerosis in hypercholesterolemia. Arterioscler Thromb Vasc Biol. 2006 Nov;26(11):2530-5. doi: 10.1161/01.ATV.0000243941.72375.15. Epub 2006 Aug 31. PMID 16946129
- [Background] Pirro M, Schillaci G, Bagaglia F, Menecali C, Paltriccia R, Mannarino MR, Capanni M, Velardi A, Mannarino E. Microparticles derived from endothelial progenitor cells in patients at different cardiovascular risk. Atherosclerosis. 2008 Apr;197(2):757-67. doi: 10.1016/j.atherosclerosis.2007.07.012. Epub 2007 Aug 27. PMID 17720166
- [Background] Affuso F, Ruvolo A, Micillo F, Sacca L, Fazio S. Effects of a nutraceutical combination (berberine, red yeast rice and policosanols) on lipid levels and endothelial function randomized, double-blind, placebo-controlled study. Nutr Metab Cardiovasc Dis. 2010 Nov;20(9):656-61. doi: 10.1016/j.numecd.2009.05.017. Epub 2009 Aug 20. PMID 19699071